CLINICAL TRIAL: NCT02464917
Title: Supplemental Oxygen Study
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Michael Nageotte, Maternal Fetal Medicine Division Director, MemorialCare Health System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 491-14
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Cesarean Section; Supplemental Oxygen; Umbilical Cord Gases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplemental oxygen (Experimental): Subjects in this arm will receive 10L/min via simple facemask
  Interventions: Device: Device: simple facemask to administer supplemental oxygen
- Room air (No Intervention): This control arm will receive no supplemental oxygen

INTERVENTIONS:
Device: Device: simple facemask to administer supplemental oxygen
  Arms: Supplemental oxygen

SUMMARY:
The purpose of this study is to compare umbilical cord gases in subjects receiving oxygen at 10L/min via simple facemask to subjects receiving room air in those presenting for scheduled cesarean sections.

DETAILED DESCRIPTION:
Objective:

To compare umbilical cord gases in subjects receiving oxygen at 10L/min via simple facemask to subjects receiving room air in those presenting for scheduled cesarean sections. The investigators hypothesize that umbilical artery pH levels will not be significantly lowered in the oxygenated group.

Primary outcome: umbilical artery pH levels in the oxygenated versus room air group

Secondary outcomes: Apgars, respiratory distress syndrome, necrotizing enterocolitis, interventricular hemorrhage, intubation, number of NICU days and neonatal mortality.

Methods:

Only term elective c-sections will be approached for study consent. Once enrolled subjects will be randomized either receive 10L/min via simple facemask or to room air. Once regional anesthesia is completed, then the facemask with oxygen will be placed. The time from oxygen administration to uterine incision will be at least 10 min. At the time of delivery umbilical cord gases will be collected by and will be processed within one hour of delivery.

Inclusion criteria:

* 18 years or older
* Scheduled cesarean section
* Singleton
* Term gestation; at 37 0/7 weeks gestation or greater

Exclusion criteria:

* Maternal lung disease including asthma
* Evidence of hypoxemia prior to enrollment
* Intrauterine growth restriction
* Chronic hypertension
* Preeclampsia
* Fetal anomalies
* Breech position
* Multiple Gestation

Statistical analysis:

Subjects will be randomized via block randomization. The estimated umbilical arterial pH in the scheduled cesarean section room air group is 7.31. To identify a 0.05 or greater difference between the control and treatment group, a power of 0.8, alpha of 0.05 the investigators would need 64 subjects total. To account for drop out the investigators intend to enroll a total of 70 subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Scheduled cesarean section
* Singleton
* Term gestation

Exclusion Criteria:

* Maternal lung disease including asthma
* Evidence of hypoxemia prior to enrollment
* Intrauterine growth restriction
* Chronic hypertension
* Preeclampsia
* Fetal anomalies
* Breech position
* Multiple gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nageotte, MD, Principal Investigator — MemorialCare Health System
Locations (1):
- Long Beach Memorial Care Center for Women at Miller Children's Hospital Long Beach and Long Beach Memorial Hospital, Long Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Supplemental Oxygen: Subjects in this arm will receive 10L/min via simple facemask
  Device: simple facemask to administer supplemental oxygen
Period: Overall Study
Arm/Group | Supplemental Oxygen | Room Air
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of participants in each groups is 35. However in supplemental oxygen group only 33 analyzed (n=2 umbilical arterial blood gas values unavailable) and in the room air group only 32 analyzed (n=1 umbilical venous blood gas value unavailable, n=1 umbilical venous and arterial blood gas value unavailable, n=1 less than 37 weeks enrolled)
Groups:
- Total: Total of all reporting groups
Arm/Group | Supplemental Oxygen | Room Air | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Overall number of participants in each groups is 35. However in supplemental oxygen group only 33 analyzed (n=2 umbilical arterial blood gas values unavailable) and in the room air group only 32 analyzed (n=1 umbilical venous blood gas value unavailable, n=1 umbilical venous and arterial blood gas value unavailable, n=1 less than 37 weeks enrolled)
  years | 33 [28.5 to 37] | 31 [26.3 to 39.5] | 32 [27.5 to 35.5]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Overall number of participants in each groups is 35. However in supplemental oxygen group only 33 analyzed (n=2 umbilical arterial blood gas values unavailable) and in the room air group only 32 analyzed (n=1 umbilical venous blood gas value unavailable, n=1 umbilical venous and arterial blood gas value unavailable, n=1 less than 37 weeks enrolled)
  Participants
    Female | 33 | 32 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Overall number of participants in each groups is 35. However in supplemental oxygen group only 33 analyzed (n=2 umbilical arterial blood gas values unavailable) and in the room air group only 32 analyzed (n=1 umbilical venous blood gas value unavailable, n=1 umbilical venous and arterial blood gas value unavailable, n=1 less than 37 weeks enrolled)
  Participants
    Caucasian | 5 | 6 | 11
    Black | 6 | 8 | 14
    Hispanic | 16 | 11 | 27
    Asian | 6 | 6 | 12
    Other / unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Umbilical Cord pH Levels
Description: marker for metabolic acidosis
Time Frame: collected at the time of delivery and all umbilical cord values resulted within 1 hour of collection
Measure: Median (Inter-Quartile Range); unit: pH
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
pH | 7.29 [7.26 to 7.3] | 7.28 [7.25 to 7.30]

2. Secondary Outcome: Umbilical Cord Base Excess
Description: marker for metabolic acidosis
Time Frame: collected at the time of delivery and all umbilical cord values resulted within 1 hour of collection
Measure: Median (Inter-Quartile Range); unit: mEq/L
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
mEq/L | -1.3 [-2.1 to -0.45] | -1.6 [-3.0 to -0.4]

3. Secondary Outcome: Umbilical Cord Partial Pressure Carbon Dioxide (pCO2)
Description: marker for metabolic acidosis
Time Frame: collected at the time of delivery and all umbilical cord values resulted within 1 hour of collection
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
mmHg | 58 [51 to 61.5] | 58 [51 to 61.5]

4. Secondary Outcome: Umbilical Cord Bicarbonate (HCO3)
Description: marker for metabolic acidosis
Time Frame: collected at the time of delivery and all umbilical cord values resulted within 1 hour of collection
Measure: Median (Inter-Quartile Range); unit: mEq/L
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
mEq/L | 26 [25 to 27] | 26 [25 to 27]

5. Secondary Outcome: Number of Newborns With an Apgar Score <7
Description: quick test performed on all babies once born that access how babies transition after birth. The following signs are given values of 0, 1, or 2 and added to compute the Apgar score. The higher the points the better. maximum points is 10. minimum score is 0. Signs: Color (0=blue/pale, 1=acrocyanotic, 2=completely pink), Heart rate (0=absent, 1=<100 minute, 2=>100 minute), Reflex irritability(0=no response, 1=grimace, 2=cry), muscle tone (0=limp, 1=some flexion, 2=active motion), Respiration (0=absent, 1=weak cry; hypoventilation, 2=good, crying)
Time Frame: completed at 5 minutes of life, Apgar <7
Measure: Number; unit: newborns
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
newborns | 0 | 0

6. Secondary Outcome: Number of Newborns With Respiratory Distress Syndrome
Description: syndrome typically affecting premature babies due to immature lung maturation or development
Time Frame: completed once infant is discharged home; anticipate 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

7. Secondary Outcome: Number of Newborns With Necrotizing Enterocolitis
Description: condition that affects newborn bowels where the tissue undergoes necrosis
Time Frame: completed once infant is discharged home; anticipate 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

8. Secondary Outcome: Number of Newborns With Intraventricular Hemorrhage
Description: condition that causes bleeding within the brain typically affecting premature babies
Time Frame: completed once infant is discharged home; anticipate 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

9. Secondary Outcome: Number of Newborns Requiring Intubation
Description: needing supplemental oxygen for the newborn through breathing device
Time Frame: completed once infant is discharged home; anticipate 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

10. Secondary Outcome: Number of Newborns Admitted to the NICU (Neonatal Intensive Care Unit)
Description: if newborns need higher intensity of care they are transferred to the Neonatal Intensive Care Unit.
Time Frame: completed once infant is discharged home; anticipate 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

11. Secondary Outcome: Neonatal Mortality
Time Frame: completed once infant is discharged home; anticipate 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen | Room Air
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Supplemental Oxygen | Room Air
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes